CLINICAL TRIAL: NCT04397718
Title: Hormonal Intervention for the Treatment in Veterans With COVID-19 Requiring Hospitalization (HITCH): A Multicenter, Phase 2 Randomized Controlled Trial of Best Supportive Care (BSC) vs BSC Plus Degarelix
Brief Title: Hormonal Intervention for the Treatment in Veterans With COVID-19 Requiring Hospitalization
Acronym: HITCH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COVID19-8900-15
Record Dates: First submitted 2020-05-14; First posted 2020-05-21 (Actual); Results first posted 2022-06-06 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo + BSC (Placebo Comparator): No active, only placebo (2 - prefilled syringes containing 3 ml of 0.9% saline) plus best supportive care.
  Interventions: Other: Saline
- Degarelix + BSC (Experimental): Active Degarelix (2 - prefilled syringes containing 3 ml of reconstituted Degarelix concentrated to 40mg/ml) plus best supportive care.
  Interventions: Drug: Degarelix

INTERVENTIONS:
Drug: Degarelix — Degarelix is an FDA-approved drug for prostate cancer
  Arms: Degarelix + BSC
Other: Saline — 09% Saline
  Arms: Placebo + BSC

SUMMARY:
The purpose of this study is to determine if temporary androgen suppression improves the clinical outcomes of Veterans who are hospitalized to an acute care ward due to COVID-19.

DETAILED DESCRIPTION:
A novel coronavirus, now termed Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2), arose late in 2019. The first confirmed cases occurred in December in Wuhan, Hubei province, China. It now infects people on six continents, spreading person to person. The World Health Organization (WHO) classified it as a global pandemic on March 11, 2020. As of April 6, 2020, there are more than 1.2 million confirmed cases and more than 70,000 deaths attributed to this virus. Every person on Earth, as well as every United States Veteran, is at risk. This is the emergent public health threat of our time.

SARS-CoV-2 is a singled stranded RNA virus related to severe acute respiratory syndrome-related coronavirus (SARS-CoV-1). SARS-CoV-2 is thought to be transmissible largely by respiratory droplets or direct contact, but might also be transmitted through aerosolization. SARS-CoV-2 disease severity ranges from no to minimal symptoms, mildly symptomatic with cough and dyspnea, to severe respiratory distress with multi-organ failure requiring admission to an intensive care unit and emergent ventilator support. Although data are evolving, the severity of illness varies with age, co-existing comorbidities, and biological sex, with older age, people with pre-existing cardiovascular disease, and males manifesting greater disease severity.

A worldwide effort is in place to contain and suppress human-to-human transmission. These public-health strategies aim to slow the rate of spread and reduce the burden on critical care infrastructure. However, there is also a need effective therapeutics. Vaccine trials are underway but potential approvals are at least a year away. Development of new drugs de novo to treat SARS2-CoV-2 will likely take even longer. Thus, the most expedient therapeutic strategy to confront this pandemic will repurpose existing FDA-approved therapeutics. One potential strategy targets viral components directly, using existing antivirals and anti-infectives currently used for other diseases. Such efforts include trials of hydroxychloroquine, remdesivir, and ribavirin. Another strategy involves targeting the human proteins, rather than viral proteins, required for SARS CoV-2 entry and replication.

ELIGIBILITY:
Inclusion Criteria:

* Male Veterans admitted to a VA hospital.
* Age > 18
* Hospitalized on an acute care ward with a diagnosis of COVID-19 contributing to hospitalization.
* Positive RT-PCR assay for SARS-CoV-2 on a nasopharyngeal swab sample.
* Severity of illness of level 3, 4 or 5 on the influenza severity scale (see Appendix A) at the time of randomization.
* The subject (or legally acceptable representative if applicable) must provide written informed consent for the trial.

Exclusion Criteria:

* History of severe hypersensitivity to degarelix or any component of their respective formulation.
* History of congenital long QT syndrome or known history of prolonged QT interval corrected by the Fridericia correction formula (QTcF) > 500 msec on electrocardiogram performed at screening.
* Planned discharge within 24 hours of treatment initiation.
* Subject is planning to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment.
* Ongoing usage of a Class IA or Class III antiarrhythmic agent. At least 5 half lives must elapse since any prior use of a Class IA or III antiarrhythmic agent prior to administration of study drug.

  --Baseline electrolyte abnormalities of Grade 3 or higher (based on CTCAE v5.0 criteria). Patients may be included if baseline electrolyte abnormalities are corrected to Grade 2 or lower prior to study drug administration.
* Myocardial infarction in the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) Class III or IV heart disease.
* Enrollment in another investigational study within 30 days of Day 1.
* Known psychiatric or substance abuse disorder that would interfere with the requirements of the trial.
* Child-Pugh Class C liver disease.
* Use of any of the following hormonal agents within Day 1 of treatment:

  1. Androgen receptor antagonists or agonists within 4 weeks,
  2. Ketoconazole or abiraterone acetate within 2 weeks,
  3. Estrogens or progestins within 2 weeks,
  4. Herbal products that contain hormonally active agents within 2 weeks.
* Unwilling or unable to comply with the study protocol.
* Any condition, which in the opinion of the investigator, would preclude participation in the trial.

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew B. Rettig, MD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (14):
- United States (14):
  - Phoenix VA Health Care System, Phoenix, AZ, Phoenix, Arizona
  - Central Arkansas VHS John L. McClellan Memorial Veterans Hospital, Little Rock, AR, Little Rock, Arkansas
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, Los Angeles, California
  - Miami VA Healthcare System, Miami, FL, Miami, Florida
  - St. Louis VA Medical Center John Cochran Division, St. Louis, MO, St Louis, Missouri
  - Brooklyn Campus of the VA NY Harbor Healthcare System, Brooklyn, NY, Brooklyn, New York
  - Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY, New York, New York
  - Philadelphia MultiService Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina
  - Memphis VA Medical Center, Memphis, TN, Memphis, Tennessee
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nickols NG, Mi Z, DeMatt E, Biswas K, Clise CE, Huggins JT, Maraka S, Ambrogini E, Mirsaeidi MS, Levin ER, Becker DJ, Makarov DV, Adorno Febles V, Belligund PM, Al-Ajam M, Muthiah MP, Montgomery RB, Robinson KW, Wong YN, Bedimo RJ, Villareal RC, Aguayo SM, Schoen MW, Goetz MB, Graber CJ, Bhattacharya D, Soo Hoo G, Orshansky G, Norman LE, Tran S, Ghayouri L, Tsai S, Geelhoed M, Rettig MB. Effect of Androgen Suppression on Clinical Outcomes in Hospitalized Men With COVID-19: The HITCH Randomized Clinical Trial. JAMA Netw Open. 2022 Apr 1;5(4):e227852. doi: 10.1001/jamanetworkopen.2022.7852. PMID 35438754
- [Derived] Nickols NG, Goetz MB, Graber CJ, Bhattacharya D, Soo Hoo G, Might M, Goldstein DB, Wang X, Ramoni R, Myrie K, Tran S, Ghayouri L, Tsai S, Geelhoed M, Makarov D, Becker DJ, Tsay JC, Diamond M, George A, Al-Ajam M, Belligund P, Montgomery RB, Mostaghel EA, Sulpizio C, Mi Z, Dematt E, Tadalan J, Norman LE, Briones D, Clise CE, Taylor ZW, Huminik JR, Biswas K, Rettig MB. Hormonal intervention for the treatment of veterans with COVID-19 requiring hospitalization (HITCH): a multicenter, phase 2 randomized controlled trial of best supportive care vs best supportive care plus degarelix: study protocol for a randomized controlled trial. Trials. 2021 Jul 5;22(1):431. doi: 10.1186/s13063-021-05389-0. PMID 34225789

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo + BSC | Degarelix + BSC
Started | 34 | 62
Completed | 27 | 47
Not Completed | 7 | 15
Not completed — Death | 7 | 11
Not completed — Lost to Follow-up | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + BSC | Degarelix + BSC | Total
Number analyzed (Participants) | 34 | 62 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (8.18) | 68.8 (8.6) | 68.5 (8.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 34 | 62 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 12 | 14
  Not Hispanic or Latino | 32 | 48 | 80
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 15 | 23 | 38
  White | 17 | 28 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 7 | 9

OUTCOME MEASURES:

1. Primary Outcome: Composite of Mortality, Ongoing Need for Hospitalization, or Mechanical Ventilation at Day 15
Description: Number of Patients who died, had a ongoing need for hospitalization, or was placed on mechanical ventilation at Day 15.
Time Frame: 15 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + BSC | Degarelix + BSC
Number analyzed (Participants) | 34 | 62
Participants | 9 | 19
Statistical Analysis 1: Comparison: Placebo + BSC vs Degarelix + BSC; Test type: Superiority; p = 0.667, Chi-squared; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.46 to 3.06] — Logistic regression adjusted for age, hypertension, and COPD

2. Secondary Outcome: Time to Clinical Improvement
Description: Time to clinical improvement as defined by a decline of 2 categories or more from the baseline modified 7-category ordinal scale of clinical status of hospitalized influenza patients or hospital discharge, whichever comes first. Participants whose condition worsened, who died, or who withdrew from the study without clinical improvement were censored. The 7-categories were defined as: 1: Not hospitalized with resumption of normal activities; 2: Not hospitalized, but unable to resume normal activities; 3: Hospitalization, not requiring supplemental oxygen; 4: Hospitalization, requiring supplemental oxygen; 5: Hospitalization, requiring nasal high-flow oxygen therapy and/or noninvasive mechanical ventilation; 6: Hospitalization, requiring extracorporeal membrane oxygenation and/or invasive mechanical ventilation; 7: Death.
Time Frame: Through discharge (an average of 8 days with a maximum of 2.5 months)
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Placebo + BSC | Degarelix + BSC
Number analyzed (Participants) | 34 | 62
Days | 5.50 [5 to 15] | 7.00 [4 to 15]
Statistical Analysis 1: Comparison: Placebo + BSC vs Degarelix + BSC; Test type: Superiority; p = 0.876, Log Rank; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.58 to 1.49] — Cox regression model adjusted for age, hypertension, and COPD

3. Secondary Outcome: Inpatient Mortality
Description: Number of patients who died during their hospital stay
Time Frame: Through discharge (an average of 8 days with a maximum of 2.5 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + BSC | Degarelix + BSC
Number analyzed (Participants) | 34 | 62
Participants | 6 | 11
Statistical Analysis 1: Comparison: Placebo + BSC vs Degarelix + BSC; Test type: Superiority; p = 0.991, Chi-squared; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.31 to 2.92] — Logistic regression adjusted for age, hypertension, and COPD

4. Secondary Outcome: Duration of Hospitalization
Description: Length of hospital stay (randomization to discharge)
Time Frame: Through discharge (an average of 8 days with a maximum of 2.5 months)
Population: Patients who died during the hospital stay were excluded.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Placebo + BSC | Degarelix + BSC
Number analyzed (Participants) | 28 | 51
Days | 5.00 [5 to 8] | 6.00 [3 to 9]
Statistical Analysis 1: Comparison: Placebo + BSC vs Degarelix + BSC; Test type: Superiority; p = 0.841, Wilcoxon (Mann-Whitney); Quantile Regression = 0, 95% CI 2-sided [-2.03 to 4.11] — Adjusted for age, hypertension, and COPD

5. Secondary Outcome: Duration of Intubation
Description: Length of time on mechanical ventilation. Length of mechanical ventilation imputed to maximum length (50 days) for patients who died on mechanical ventilation or who were on mechanical ventilation, but date removed was unknown. Length of mechanical ventilation imputed to 0 for patients never on mechanical ventilation.
Time Frame: Through discharge (an average of 8 days with a maximum of 2.5 months)
Population: Patients who died and who were not on mechanical ventilation prior to death were excluded (N=4).
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Placebo + BSC | Degarelix + BSC
Number analyzed (Participants) | 33 | 59
Days | 0.00 [0 to 0] | 0.00 [0 to 0]
Statistical Analysis 1: Comparison: Placebo + BSC vs Degarelix + BSC; Test type: Superiority; p = 0.746, Wilcoxon (Mann-Whitney); Quantile Regression = 0, 95% CI 2-sided [0 to 0] — Adjusted for age, hypertension, and COPD

6. Secondary Outcome: Time to Normalization of Temperature.
Description: Length of time for temperature to be less than < 37.5 degree Celsius for 48 hours
Time Frame: Through discharge (an average of 8 days with a maximum of 2.5 months)
Population: Patients with a fever (temperature greater than or equal to 37.5 degrees Celsius) at baseline.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Placebo + BSC | Degarelix + BSC
Number analyzed (Participants) | 7 | 17
Days | 5.00 [2 to 18] | 3.00 [1 to 3]
Statistical Analysis 1: Comparison: Placebo + BSC vs Degarelix + BSC; Test type: Superiority; p = 0.1, Log Rank; Hazard Ratio (HR) = 2.3, 95% CI 2-sided [0.72 to 7.39] — Cox regression model adjusted for age, hypertension, and COPD

7. Secondary Outcome: Maximum Severity of COVID19 Illness.
Description: Maximum severity score on the modified 7-category ordinal scale of clinical status of hospitalized influenza patients. The 7-categories were defined as: 1: Not hospitalized with resumption of normal activities; 2: Not hospitalized, but unable to resume normal activities; 3: Hospitalization, not requiring supplemental oxygen; 4: Hospitalization, requiring supplemental oxygen; 5: Hospitalization, requiring nasal high-flow oxygen therapy and/or noninvasive mechanical ventilation; 6: Hospitalization, requiring extracorporeal membrane oxygenation and/or invasive mechanical ventilation; 7: Death.
Time Frame: Through discharge (an average of 8 days with a maximum of 2.5 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + BSC | Degarelix + BSC
Number analyzed (Participants) | 34 | 62
Participants
  Hospitalization, not requiring supplemental oxygen | 4 | 8
  Hospitalization, requiring supplemental oxygen | 20 | 26
  Hospitalization,req. nasal high-flow oxygen therapy &/or noninvasive mechanical ventilation | 4 | 14
  Hospitalization, req. extracorporeal membrane oxygenation &/or invasive mech. ventilation | 0 | 3
  Death | 6 | 11
Statistical Analysis 1: Comparison: Placebo + BSC vs Degarelix + BSC; Test type: Superiority; p = 0.425, Fisher Exact; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.33 to 2]; Logistical regression adjusted for age, hypertension, COPD, and baseline severity score

8. Secondary Outcome: Composite of Mortality, Ongoing Need for Hospitalization, or Mechanical Ventilation at Day 30
Description: Number of Patients who died, had a ongoing need for hospitalization, or was placed on mechanical ventilation at Day 30.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + BSC | Degarelix + BSC
Number analyzed (Participants) | 34 | 62
Participants | 7 | 15
Statistical Analysis 1: Comparison: Placebo + BSC vs Degarelix + BSC; Test type: Superiority; p = 0.688, Chi-squared; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.44 to 3.42] — Logistic regression adjusted for age, hypertension, and COPD

ADVERSE EVENTS:
Time Frame: From randomization through day 60.
Description: AE and SAE data were collected through spontaneous local SC/LSI/Co-I contact, during in-person study visits, and gathered during telephone contacts and medical record reviews when performed.
Arm/Group | Placebo + BSC | Degarelix + BSC
All-Cause Mortality (participants affected / at risk) | 7/34 | 11/62
Serious Adverse Events (participants affected / at risk) | 11/34 | 19/62
Other Adverse Events (participants affected / at risk) | 8/34 | 13/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + BSC (N=34) | Degarelix + BSC (N=62)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 3 (3)
COVID-19 pneumonia (Infections and infestations) | 4 (4) | 5 (5)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
SARS-CoV-2 sepsis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Mouth haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + BSC (N=34) | Degarelix + BSC (N=62)
Accelerated idioventricular rhythm (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Injection site pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injection site reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tooth avulsion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Hot flush (Vascular disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/18/NCT04397718/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-05): https://cdn.clinicaltrials.gov/large-docs/18/NCT04397718/SAP_001.pdf